CLINICAL TRIAL: NCT00331032
Title: An Expanded Phase I Randomized Placebo Controlled Trial of the Safety and Tolerability of 3 Percent w/w SPL7013 Gel (VivaGel™) in Healthy Young Women When Administered Twice Daily for 14 Days
Brief Title: VivaGel™ in Healthy Young Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 05-0121; SPL7013-004
Record Dates: First submitted 2006-05-25; First posted 2006-05-29 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Herpes Simplex II
Keywords: VivaGel™, sexually transmitted, microbicide, herpes simplex
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1: 3% w/w SPL7013 Gel (Experimental): 40 subjects VivaGel™.
  Interventions: Drug: 3% w/w SPL7013 Gel
- 2: Placebo (Placebo Comparator): 20 subjects placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 3% w/w SPL7013 Gel — Twice-daily vaginal application of 3.5 g of VivaGel™ (Carbopol®-based gel with 3% w/w SPL7013) in single use pre-filled applicators.
  Arms: 1: 3% w/w SPL7013 Gel
Drug: Placebo — Placebo gel (Carbopol®-based formulation alone) in single use pre-filled applicators.
  Arms: 2: Placebo

SUMMARY:
The purpose of this study is to test the safety and tolerability of a medication applied vaginally twice daily in females versus placebo (inactive substance). Study participants will include 60 women, ages 18-24, non-pregnant, previously sexually active, Human Immunodeficiency Virus (HIV) negative and sexually transmitted infection (STI) free, in San Francisco or Kisuma, Kenya. Each study participant will be followed for 14 days of product use and an additional 7 days for safety assessments. Study procedures will include a physical exam with a pap smear, urine testing, blood sample testing, and a colposcopy (exam of the vagina and cervix using a lighted magnifying instrument). Information learned from this study may help to develop a safe and effective medication that could prevent herpes simplex virus and HIV. Participants may be involved in study related procedures for up to 55 days.

DETAILED DESCRIPTION:
Over half of global human immunodeficiency virus (HIV) infections occur among those aged 18-24 years and young women are at a particularly high risk of acquiring genital herpes caused by herpes simplex virus type 2 (HSV-2) and other sexually transmitted infections (STI). This is a phase I, randomized, double blind, clinical trial of twice-daily vaginal VivaGel™ (n equals 40) versus placebo gel (n equals 20). The primary aim of this protocol is to test the safety and tolerability of VivaGel™ in young women, with the long-term aim of testing the efficacy of this compound in preventing HSV-2 in a future phase II/III trial. A total of 60 young women aged 18-24, non-pregnant, previously sexually active, STI and HIV free, in San Francisco and in Kisumu, Kenya will participate in this study. Eligibility screening will include medical history, pelvic exam with a Pap smear, urine pregnancy testing, HIV and STI counseling and testing, hematology testing and liver and renal function testing. Eligible participants will undergo a pelvic exam with colposcopy. Vaginal swabs will be collected to evaluate H2O2-producing lactobacilli and Gram stain, Chlamydia, gonorrhea, and prostate specific antigen (PSA) (to confirm lack of exposure to semen). Endocervical samples will be collected to measure immunological status. Blood will be collected to conduct hematology and liver and renal function testing, and plasma will be collected and stored for batch testing. Subjects will be provided with the investigational product or placebo, given a Daily Study Record, instructed how to use the product, complete the Daily Study Record, and report any adverse events (AEs). Follow-up visits will occur on Days 2, 7, 14, and 21. The primary study objective will be to determine the safety and tolerability of VivaGel™ applied vaginally twice daily for 14 days in HIV negative and STI-free young women. Safety assessments, comparing the VivaGel™ group to the placebo gel group, will include: incidence and severity of AEs, including genital tract signs and symptoms and mucosal changes as observed by colposcopy; vaginal microflora, including colonization with H2O2-producing lactobacilli; and laboratory parameters, including serum chemistry and hematology. The tolerability assessment, comparing the VivaGel™ group to the placebo gel group will include the proportion of participants who discontinued product use due to overt (i.e. observable) AEs, ascertained through a standardized questionnaire. The secondary objective of the study will be to report the effect of VivaGel™ applied vaginally twice daily for 14 days on the immune microenvironment in the lower genital tract of young women. Specifically, this will be tested by determining its effect on: the number and activation levels of endocervical immune cell populations; Secretory Leukocyte Protease Inhibitor (SLPI) levels; innate mucosal defenses, including local levels of cytokines in cervical secretions, and Toll-Like Receptor (TLR) expression by cervical immune cells; and the presence and expression levels of the HIV co-receptors CCR5 and CXCR4, and of their principal chemokine ligands by endocervical immune cells.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily given written informed consent to participate in the study.
* Subject is female and aged between 18 and 24 years, inclusive.
* Subject is sexually active.
* Subject should have a menstrual cycle length of at least 25 days.
* Subject is in good health, as determined by medical history, a baseline physical examination, and clinical laboratory tests.
* Subject agrees to comply with all study procedures.
* Subject has no significant abnormal vaginal microflora (abnormal flora defined as Nugent score greater than or equal to 7) at screening.
* Subject has a negative urine pregnancy test at screening and enrollment.
* Participant must agree to abstain from all sexual activities involving intercourse or other forms of vaginal penetration 7 days prior to the Enrollment Visit through the completion of all follow-up visits and procedures.

Exclusion Criteria:

* Subject has received or is anticipated to receive a new prescription systemic or topical medication within 14 days prior to the start of dosing. Subjects may be enrolled if stable on existing therapy as determined by the Principal Investigator.
* Subject has received any new long-acting treatments [e.g. depot formulation including medroxyprogesterone acetate (DMPA) form of hormonal birth control]. Subjects may be enrolled if stable (greater than 3 months) on existing therapy as determined by the Principal Investigator.
* Subject has received an investigational drug within 30 days or 10 half-lives of the drug, whichever is longer, prior to entering this study, or is planning to receive another investigational drug while participating in this study.
* Subject has a history of significant drug allergy.
* Subject has a history of latex allergy.
* Biological and hematological parameters are outside of the laboratory's normal reference ranges. Subjects with grade 1 laboratory abnormalities can be included if the Principal Investigator judges that the deviations are not clinically relevant.
* Subject has a clinically significant history of systemic allergic disease (e.g., clinically significant urticaria, clinically significant atopic dermatitis).
* Subject has a history of recurrent vaginal infections, irritation or localized reaction to vaginally applied agents.
* Subject has an unpredictable or irregular menstrual cycle that will not allow scheduling of the colposcopic examinations outside menstruation as required for the protocol.
* Subject has a recent (within 3 months) history of intermenstrual bleeding.
* Subject has an active, uncontrolled medical condition (e.g., neurological, gastrointestinal, renal, hepatic, cardiovascular, pulmonary, metabolic, endocrine, hematological, genitourinary or other major disorder), or psychiatric illness (e.g., depression, schizophrenia).
* Subject had a clinically significant illness within 30 days prior to screening.
* Subject has used a vaginal preparation within 30 days prior to screening.
* Subject has a clinically detectable genital abnormality (i.e. vulvar, vaginal, cervical, perianal ulcer and/or deep epithelial disruption).
* Subject has signs, as seen on pelvic exam, consistent with an Sexually Transmitted Infection (STI), other genital tract infection - other than bacterial vaginosis (BV) - or trauma, including but not limited to: vaginitis, cervicitis, and laboratory findings indicative of genital tract infection other than asymptomatic BV.

Note: Signs of asymptomatic BV include the presence of white to grey homogeneous discharge, positive whiff test (amine odor) with addition of KOH, pH>4.5, presence of clue cells, decrease in lactobacilli morphotypes, and increase in non-lactobacilli morphotypes. Women with clinical or gram stain evidence of BV and symptoms (discharge, odor, itching), or yeast colonization and symptoms at screening should be treated and re-evaluated for inclusion. Women without BV symptoms, but who have clinical or gram stain evidence of BV, or asymptomatic yeast colonization, are eligible.

* Subject tests positive for serum antibodies to human immunodeficiency virus 1 and/or 2 (HIV-1 and/or HIV-2).
* Subject tests positive for serum antibodies to herpes simplex virus, type 2 (HSV-2).
* Subject tests positive for Chlamydia, gonorrhea, trichomonas, syphilis or a urinary tract infection at screening or enrollment.

Note: Women who have an STI or are symptomatic and have a positive urine culture (urinary tract infection - UTI) at screening will be referred for and/or given treatment. Following completion of treatment, women with a negative repeat test may be reconsidered for study participation.

* Subject has an abnormal Pap smear at screening.
* Subject has history in the last three months of: an IUD, vaginal contraceptive ring, a pregnancy, cervical cryotherapy or laser therapy, gynecologic surgery.
* Subject is currently breast feeding or is planning on breast feeding while participating in this study.
* Subject, in the opinion of the Principal Investigator, should not participate in the study.
* Women with colposcopic evidence of deep epithelial disruption at the enrollment visit will be excluded. In addition, based on the investigator's (medical examiner's) opinion any colposcopic finding or any finding (normal or abnormal) that could interfere with colposcopic examinations may also lead to exclusion. In this case, the investigator may have the subject return within the screening window to determine if the abnormality has cleared, and if she is eligible for enrollment.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2006-12; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Tolerability will assess the degree to which overt Adverse Events can be tolerated by the study participants. | Tolerability measures will be assessed at Days 2, 7, and 14 visits.
Safety will be assessed by laboratory tests and clinical Adverse Events. | Safety assessed after 2, 7, and 14 days of product use and 7 days following the completion of product use (Day 21).

SECONDARY OUTCOMES:
Presence and expression levels of Human Immunodeficiency Virus co-receptors CCR5 and CXCR4, and their principal chemokine ligands by endocervical immune cells. | Immunologic factors of the genital tract will be measured using cervicovaginal specimens collected at enrollment, Day 7, Day 14, and Day 21.
Secretory Leukocyte Protease Inhibitor levels. | Immunologic factors of the genital tract will be measured using cervicovaginal specimens collected at enrollment, Day 7, Day 14, and Day 21.
Number and activation levels of endocervical immune cell populations. | Immunologic factors of the genital tract will be measured using cervicovaginal specimens collected at enrollment, Day 7, Day 14, and Day 21.
Innate mucosal defenses, including local levels of cytokines in cervical secretions, and Toll-Like Receptor expression by cervical immune cells. | Immunologic factors of the genital tract will be measured using cervicovaginal specimens collected at enrollment, Day 7, Day 14, and Day 21.

CONTACTS AND LOCATIONS:
Locations (2):
- University of California San Francisco, San Francisco, California, United States
- Kenya Medical Research Institute, Kisumu, Kenya

REFERENCES:
- [Result] Cohen CR, Brown J, Moscicki AB, Bukusi EA, Paull JR, Price CF, Shiboski S. A phase I randomized placebo controlled trial of the safety of 3% SPL7013 Gel (VivaGel(R)) in healthy young women administered twice daily for 14 days. PLoS One. 2011 Jan 20;6(1):e16258. doi: 10.1371/journal.pone.0016258. PMID 21311578